CLINICAL TRIAL: NCT02270255
Title: Prospective Blinded Study Looking at PO/IV Analgesia Alone Versus PO/IV Analgesia With Superior Hypogastric Nerve Block for Uterine Artery Embolization Pain Management
Brief Title: Superior Hypogastric Nerve Block for Pain Control Post-uterine Fibroid Embolization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Louis-martin Boucher, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4242
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Leiomyoma
Keywords: embolization; analgesia
MeSH Terms: conditions — Leiomyoma; Agnosia | interventions — Ropivacaine; Injections, Subcutaneous; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Sham Comparator): Sham procedure. Subcutaneous injection of 5cc of 1% Xylocaine in the periumbilical region.
  Interventions: Procedure: Subcutaneous injection; Drug: 1% Xylocaine
- Sup Hypogastric Nerve block group (Experimental): Superior hypogastric nerve block performed during UFE. 20cc of 0.75% Ropivacaine injected at the superior hypogastric nerve plexus.
  Interventions: Procedure: Superior hypogastric nerve block; Drug: 0.75% Ropivacaine

INTERVENTIONS:
Procedure: Superior hypogastric nerve block — 21g Chiba needle advanced into the superior hypogastric plexus via an anterior infraumbilical approach using the arterial catheter as a fluoroscopic landmark to target the vertebral body below.
  Arms: Sup Hypogastric Nerve block group
Drug: 0.75% Ropivacaine — 20 ml of 0.75% Ropivacaine
  Other Names: Naropin
  Arms: Sup Hypogastric Nerve block group
Procedure: Subcutaneous injection — Injection into subcutaneous tissues in periumbilical region
  Arms: Control group
Drug: 1% Xylocaine — 5ml of 1% Xylocaine
  Other Names: Lidocaine
  Arms: Control group

SUMMARY:
Uterine fibroid embolization (UFE) is now an accepted treatment of uterine fibroids. However the procedure is often very painful and, in many centres, patients are admitted overnight with patient controlled analgesic (PCA) pumps for pain control and discharged the next day with heavy pain medications. The goal of this study is to evaluate the effectiveness of a superior hypogastric nerve block (SHGNB) in controlling the pain post-UFE.

DETAILED DESCRIPTION:
This is a double blinded study in which the patients and the primary operators of the UFE as well as the post-procedural caregivers are blinded to whether the patients have received a sham procedure (injection of xylocaine in the skin in the peri-umbilical region) or the superior hypogastric nerve block.

The superior hypogastric nerve block (SHGNB) consists of advancing a 21g Chiba needle via an anterior approach up to the superior hypogastric nerve plexus and injecting 20cc of 0.75% Ropivacaine which is a long lasting local anesthetic agent. The nerve plexus is positioned below the aortic bifurcation along the anterior surface of the vertebral body. By fluoroscopy, the location can be identified by having a catheter crossing the aortic bifurcation. That way, we are able to target, under fluoroscopy, the anterior surface of the vertebral body just below the catheter.

Our UFE starts with a right common femoral artery (CFA) access. The catheter is crossed to the left side and the left uterine artery embolized with polyvinyl alcohol (PVA) 500-700 particles. The operator will then leave the room. Another operator will come and perform either the hypogastric nerve block or the sham procedure (injection of xylocaine in the periumbilical subcutaneous tissues). If the hypogastric nerve block is done, the needle is advanced into position via an anterior periumbilical approach under fluoroscopic guidance. Once the bony surface is contacted, 3 cc of xylocaine is injected to numb the area and then 3-6 cc of contrast is injected to ensure that it drapes the anterior vertebral body surface. If it spreads along both sides of the vertebral body and there is no vascular intravasation of contrast, the 20 cc of Ropivacaine is injected. If it only drapes one side, 10 cc is injected and the needle repositioned to the other side, the position verified with contrast, and the left over 10 cc of Ropivacaine injected.

After the block or sham procedure is done, the primary operator enters the room again and the UFE completed with embolization of the right uterine artery.

The patient is transferred to the recovery room and monitored. Pain medication including fentanyl and midazolam are offered at routine interval or on patient request. Pain scales are measured routinely and the patient is discharge home with a pain survey with visual analog pain scales to be performed routinely for 10 days.

The patient is followed up in 4-6 months with a follow-up magnetic resonance imaging (MRI) and consultation to look at the results of the procedure.

Comparison of the pain scale reports and use of pain medication will be evaluated between both groups to determine if there is a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. All women with symptomatic fibroids or adenomyosis that have requested and been approved for uterine artery embolization
2. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Patients in whom the vascular anatomy prevents access to the superior hypogastric nerve plexus safely
2. Patients who have known allergy to the anesthetic agent
3. Patients with signs of skin infection at the entry site of the needle used to place the nerve block
4. Patients with signs of infection such as fever
5. Patients with history of inflammatory bowel disease of with signs of colitis
6. Patients with uncorrectable abnormal coagulation status (INR >1.5 and plt < 50000 without use of anticoagulation agents)
7. Patients with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study.
8. Patients who are uncooperative, cannot follow instructions, or who are unlikely to comply with follow-up appointments or fill-out the post-procedural pain questionnaires.
9. Patients with a mental state that may preclude completion of the study procedure or is unable to provide informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Martin NJ Boucher, MD/PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasuli P, Jolly EE, Hammond I, French GJ, Preston R, Goulet S, Hamilton L, Tabib M. Superior hypogastric nerve block for pain control in outpatient uterine artery embolization. J Vasc Interv Radiol. 2004 Dec;15(12):1423-9. doi: 10.1097/01.RVI.0000137406.09852.A4. PMID 15590800
- [Derived] Yoon J, Valenti D, Muchantef K, Cabrera T, Toonsi F, Torres C, Bessissow A, Bandegi P, Boucher LM. Superior Hypogastric Nerve Block as Post-Uterine Artery Embolization Analgesia: A Randomized and Double-Blind Clinical Trial. Radiology. 2018 Oct;289(1):248-254. doi: 10.1148/radiol.2018172714. Epub 2018 Jul 10. PMID 29989515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2015 and February 2017, 87 patients were approached for enrollment. All patients fit the inclusion criteria, and no patients were excluded. However, 43 of the 87 patients (49%) declined participation in the study, leaving 44 patients (51%) who agreed to participate.
Pre-assignment Details: No enrolled participants were excluded from the study. Data were complete for all participants up to the time of discharge from the postanesthesia care unit (PACU). Forty-three of the 44 participants (98%) completed the home survey; one participant (2%) was lost to follow-up.
Period: Overall Study
Arm/Group | Control Group | Sup Hypogastric Nerve Block Group
Started | 22 | 22
Complete Data at Discharge PACU | 22 | 22
Complete Data From Home Survey | 21 | 22
Completed | 21 | 22
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Same as assignment population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Sup Hypogastric Nerve Block Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (5.2) | 47 (5.7) | 46.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — McGill University Health Centre
  participants
    Canada | 22 | 22 | 44
Pain sensitivity [Mean (Standard Deviation); unit: units on a scale] — Person self-evaluation of pain of vaccine on scale of 0-10/10 Visual analog scale (VAS). Patient rates pain on a scale from 0 to 10, 0 being no pain at all and 10 being the worse pain they could ever imagine.
  units on a scale | 3.2 (2.2) | 3.5 (2.3) | 3.35 (2.2)
Pain of regular menstrual cramps [Mean (Standard Deviation); unit: units on a scale] — Patients self-reporting of pain of average menstrual cramp on a scale form 0 to 10 (Visual analog scale - VAS), 0 being no pain at all and 10 being the worse pain they could ever imagine.
  units on a scale | 6.3 (2.5) | 6.9 (1.7) | 6.6 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: mg Equivalent Morphine Used Until Discharge From Recovery Room to Control Pain Level Below 4/10 (VAS)
Description: mg equivalent morphine used until discharge from recovery room to maintain pain level below 4/10 (visual analog scale 0/10=no pain to 10/10=worse pain the patient could imagine)
Time Frame: 6 hrs (from time of end of UFE to time of discharge from recovery room)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Control Group | Sup Hypogastric Nerve Block Group
Number analyzed (Participants) | 22 | 22
mg | 11 (9) | 5.1 (5.8)

2. Secondary Outcome: Number of Patients With Serious Adverse Reactions From Superior Hypogastric Nerve Block
Description: Number of patients with Grade C/D/E/F adverse events (Society of Interventional Radiology (SIR) Classification). Per Society of Interventional Radiology (SIR) Classification: Grade C, require therapy, brief hospitalization (<48 hours); Grade D, require major therapy, unplanned increased level of care, prolonged hospitalization (>48 hours); Grade E, permanent adverse sequelae; Grade F, death.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Sup Hypogastric Nerve Block Group
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 4-6 months
Description: SIR Classification definition of adverse events.
Arm/Group | Control Group | Sup Hypogastric Nerve Block Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=22) | Sup Hypogastric Nerve Block Group (N=22)
Pain during the block procedure itself (Nervous system disorders) | 0 | 6 — Temporary discomfort/pain during placement of the block needle.
Hard fibroid needing use of 18g needle (Reproductive system and breast disorders) | 0 | 1
Tachycardia, transient, from Xylocaine with epi injection (Cardiac disorders) | 0 | 1 — To ensure no intravascular injection of long-acting block agent, a test dose of Xylocaine with epi is injected. One patient had a transient tachycardia confirming intravascular uptake and needing change in needle position.
Aspiration of blood (Vascular disorders) | 0 | 1 — Aspiration of blood prior to injecting anesthetic, needing needle repositioning.
Temporary heat sensation in foot (Nervous system disorders) | 0 | 1 — Presumably from sympathetic chain blockade
Temporary heaviness in foot (Nervous system disorders) | 0 | 1 — Resolved by the end of the time in the PACU

LIMITATIONS AND CAVEATS:
Small number of patients. Single centre study. Occasional use of different narcotics needing morphine equivalent calculations. SHAM procedure did not place a needle as deep as in the study group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT02270255/Prot_SAP_000.pdf